CLINICAL TRIAL: NCT02063763
Title: Use of TPO-mimetics to Prepare for Splenectomy in Adult Patients With Primary Immune Thrombocytopenia. Brooklyn Observational Retrospective Study.
Brief Title: TPO-mimetics Before Splenectomy in Adult Primary Immune Thrombocytopenia Patients.
Acronym: ITP0614
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: ITP0614
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Adult Patients; Immune Primary Thrombocytopenia; Splenectomy; TPO-mimetics
Keywords: Adult patients; Immune primary thrombocytopenia; Splenectomy; TPO-mimetics; Eltrombopag; Romiplostim

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims at analyzing the therapeutic activity of TPO-mimetics Eltrombopag and Romiplostim as bridge therapy for splenectomy in adult patients with primary immune thrombocytopenia.

DETAILED DESCRIPTION:
Adult immune primary thrombocytopenia is an autoimmune malignancy characterized by platelet destruction and inadequate platelet production. Its incidence is of three cases per 100,000 people a year, with a prevalence in women in young and older adults.

Splenectomy is, still today, the therapeutic approach that offers a bigger guarantee of a long term response (around 60+70%). Nevertheless, splenectomy may be accompanied by peri-operative complications in almost 10% of patients, which in rare cases may be fatal. These are normally hemorrhagic complications due to low platelet count. Thus, a previous therapy to increase platelets is advisable before any splenectomy.

In patients who are refractory to corticosteroids and immunoglobulins or when its use is not indicated, splenectomy has a potential risk of more complications. Since the last few years, we count with TPO-mimetic drugs, specific for c-MPL receptor, able to stimulate platelet production, such as romiplostim and eltrombopag.

Nowadays, TPO-mimetics are allowed in Italy when patients refuse splenectomy or when splenectomy is not contraindicated, but being ITP with a low platelet count (< 20-50.000/mmc) a potential contraindication to splenectomy due to hemorrhagic events, these drugs should be considered. Nevertheless, there are no data on therapeutic risks and safety of these agents when used for this indication. The aim of the present study is to verify, on an Italian national scale, the frequency of use, its impact and the safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or chronic ITP in symtomatic phase.
* 18 years of age or older.
* Indication for splenectomy due to refractory response to a previous therapy.
* Have used eltrombopag or romiplostim to increase platelet count before splenectomy.
* Have undergone splenectomy.

Exclusion Criteria:

* No informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ITP adult patients having undergone splenectomy after a bridge therapy with eltrombopag or romiplostim.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2015-02-26 (Actual); Study Completion 2015-02-26 (Actual)

PRIMARY OUTCOMES:
Number of patients responding to TPO-mimetics | Six months.
  According to platelet count and presence or absence of hemorrhagic events.

SECONDARY OUTCOMES:
Number of patients on TPO-mimetics eltrombopag and romiplostim as bridge therapy before splenectomy. | Six months.
Frequency and ways of administration. | Six months
Number of hemorrhagic events. | At thirty days from splenectomy.
  Number and seriousness of hemorrhagic, thrombotic and infectious events at 30 days from splenectomy.
Frequency of toxicity. | Six months
  NCI CTCAE v. 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, Pr., Study Chair — Clinica Ematologica, DISM, Azienda Ospedaliera Universitaria S. M. Misericordia
Locations (14):
- Italy (14):
  - U.O.C di Ematologia P.O. "S.Giuseppe Moscati", Aversa
  - UOC Ematologia Ospedale " Mons. Dimiccoli", Barletta
  - Policlinico di Careggi, Florence
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Unità Operativa Complessa) - Medicina Generale - Sezione di Ematologia - Ospedale Versilia USL 12 Toscana, Lido di Camaiore
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Ospedale Niguarda " Ca Granda" - SC Ematologia Blocco SUD, Ponti Est, Scala E, 4° piano, Milan
  - Unità Trapianto di Midollo Ist. Nazionale Tumori, Milan
  - Azienda Ospedaliera "S.Gerardo", Monza
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - A.O. Santa Maria - Terni S.C Oncoematologia, Terni
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation — http://www.gimema.it